CLINICAL TRIAL: NCT00063986
Title: Minimally Invasive Esophagectomy (MIE): A Multicenter Feasibility Study
Brief Title: Esophagectomy in Treating Patients With High-Grade Dysplasia of the Esophagus or Stage I, Stage II, or Stage III Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000305866; U10CA021115 (NIH); E2202 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; minimally invasive esophagectomy (MIE)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minimally invasive esophagectomy (MIE) (Experimental): Within 4 weeks of registration patients will undergo minimally invasive esophagectomy (MIE). However, there will be up to 5 months allowed between registration and MIE for those patients needing neoadjuvant therapy prior to undergoing MIE.
  Interventions: Procedure: Minimally invasive esophagectomy (MIE)

INTERVENTIONS:
Procedure: Minimally invasive esophagectomy (MIE) — Within 4 weeks of registration patients will undergo minimally invasive esophagectomy (MIE). However, there will be up to 5 months allowed between registration and MIE for those patients needing neoadjuvant therapy prior to undergoing MIE.

SUMMARY:
RATIONALE: Laparoscopic-assisted surgery and video-assisted thoracoscopy are less invasive types of surgery for esophageal cancer that may have fewer side effects and improve recovery.

PURPOSE: This phase II trial is studying how well laparoscopic-assisted surgery and video-assisted thoracoscopy work in treating patients who are undergoing esophagectomy for high-grade dysplasia of the esophagus or stage I, stage II, or stage III esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of performing minimally invasive esophagectomy (MIE), in terms of 30-day mortality, in patients with high-grade dysplasia of the esophagus or stage I-III esophageal cancer.
* Determine the complications associated with this procedure in these patients.
* Determine the rate at which conversion to open operation is required in patients undergoing this procedure.
* Determine the length of the operation, duration of intensive care unit stay, and length of hospital stay in patients undergoing this procedure.
* Determine feasibility and conversion rate of MIE after neoadjuvant therapy.
* Assess the effectiveness of lymph node dissection by MIE by recording the total number of lymph nodes dissected.
* Assess outcomes at follow-up to three years.

OUTLINE: This is a multicenter study.

Patients undergo minimally invasive esophagectomy comprising video-assisted thoracoscopy to mobilize the thoracic esophagus in combination with laparoscopy to complete the esophagectomy and a neck incision to mobilize the cervical esophagus. Mortality at 30 days is assessed.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ACTUAL ACCRUAL: A total of 110 patients were accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

DISEASE CHARACTERISTICS:

* High grade dysplasia of the esophagus who would undergo esophagectomy OR esophageal cancer at stage T1-T3, N0-N1 who require esophagectomy (patients with M1 disease and/or bulky lymph node involvement were excluded).
* Pathological confirmation of a diagnosis of cancer or high-grade dysplasia of the esophagus by biopsy.
* Computerized tomography (CT) scan of chest and abdomen within 6 weeks prior to registration
* Stomach must be available for conduit
* Age of 18 and over
* ECOG performance status of 0-2
* Creatinine less than 2 mg/dL
* Patients with esophageal cancer who would be treated with neoadjuvant chemotherapy and/or radiation were eligible. If patients were registered prior to receiving neoadjuvant chemotherapy they were allowed up to 5 months to complete therapy and any restaging that was necessary before operation was performed.
* The patient was considered an appropriate candidate for surgery based on preoperative clinical staging and physiological factors prior to registration as documented in the surgical plan. Pre-operative staging should include:

  * Endoscopic ultrasound (EUS)
  * Positron emission tomography (PET) scan and/or laparoscopic staging (Laparoscopic staging could be performed on the day of resection. Additional evaluation was recommended if the PET scan suggested distant metastatic disease.)

EXCLUSION CRITERIA:

* Cancer extending into the stomach more than 20%
* Prior anti-reflux or gastric operations
* Prior right thoracotomy
* Prior major neck operation other than the removal of superficial skin lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2004-06-24 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Luketich, MD, Study Chair — University of Pittsburgh
Locations (41):
- United States (41):
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Medical City Dallas Hospital, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on March 3, 2004, accrued its first patient on June 24, 2004, and closed on August 15, 2008. A total of 110 patients were accrued for this study.
Groups:
- Minimally Invasive Esophagectomy (MIE): Within 4 weeks of registration patients will undergo minimally invasive esophagectomy (MIE). However, there will be up to 5 months allowed between registration and MIE for those patients needing neoadjuvant therapy prior to undergoing MIE.
  Only eligible and treated patients are included in the primary analysis.
Period: Overall Study
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Started | 110
Treated | 105
Eligible and Treated | 104
Completed | 104
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Ineligible | 1
Not completed — Intra-operatively ineligible | 4

BASELINE CHARACTERISTICS:
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 104
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 83
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Peri-operative Mortality at 30 Days
Description: The primary endpoint is 30-day peri-operative mortality rate. Proportion of patients died within 30 days of surgery will be reported.
Time Frame: Assessed at 30 days from surgery
Population: Eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 104
proportion of participants | 0.029 [0.008 to 0.073]

2. Secondary Outcome: Rate of Conversion to Open Operation
Description: Proportion of patients who required conversion to operation will be reported.
Time Frame: Assessed at surgery
Population: Eligible and treated patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 104
Proportion of patients | 0.087 [0.004 to 0.158]

3. Secondary Outcome: Duration of Operating Time
Description: The length of the operation (total of thoracic and abdominal components) is recorded.
Time Frame: Assessed at surgery
Population: Eligible and treated patients are included in this analysis. Out of 104 eligible and treated patients, 10 patients' length of operation data were unavailable, so the results are based on data from 94 patients.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 94
Minutes | 330 [120 to 813]

4. Secondary Outcome: Duration of Intensive Care Stay
Description: Number of post-operative days in intensive care is reported.
Time Frame: Assessed after surgery until patients are out of intensive care
Population: Eligible and treated patients are included in this analysis. Out of 104 eligible and treated patients, duration of intensive care stay is missing for 3 patients, so the results are based on data from 101 patients.
Measure: Median (Full Range); unit: Days
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 101
Days | 2 [0 to 39]

5. Secondary Outcome: Overall Length of Hospital Stay
Description: The number of days patients stayed in the hospital after surgery is reported.
Time Frame: Assessed after surgery until patients are out of hospital
Population: Eligible and treated patients are included in this analysis. Out of 104 eligible and treated patients, duration of hospital stay is missing for 3 patients, so the results are based on data from 101 patients.
Measure: Median (Full Range); unit: Days
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 101
Days | 9 [4 to 138]

6. Secondary Outcome: Total Number of Lymph Nodes Dissected
Description: The total number of lymph nodes dissected is reported to assess the effectiveness of lymph node dissection by MIE.
Time Frame: Assessed at surgery
Population: Eligible and treated patients are included in this analysis. Out of 104 eligible and treated patients, the number of lymph nodes removed is missing for 1 patient, so the results are based on data from 103 patients.
Measure: Median (Full Range); unit: Lymph nodes
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 103
Lymph nodes | 19 [2 to 55]

7. Secondary Outcome: 3-year Survival Rate
Description: Patients are followed for survival for 3 years from registration. Overall survival is defined as the time from operation to death.
Time Frame: Assessed at 3 years
Population: Eligible and treated patients are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 104
proportion of participants | 0.584 [0.477 to 0.676]

8. Secondary Outcome: 30-day Peri-operative Mortality After Neoadjuvant Therapy
Description: Proportion of patients with neoadjuvant therapy died within 30 days of operation is reported.
Time Frame: Assessed at 30 days after surgery
Population: 35 eligible and treated patients with neoadjuvant therapy are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 35
Proportion of patients | 0.057 [0.010 to 0.169]

9. Secondary Outcome: Rate of Conversion to Open Operation After Neoadjuvant Therapy
Description: Proportion of patients with neoadjuvant therapy required conversion to open operation is reported.
Time Frame: Assessed at surgery
Population: 35 eligible and treated patients with neoadjuvant therapy are included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Number analyzed (Participants) | 35
Proportion of patients | 0.086 [0.018 to 0.231]

ADVERSE EVENTS:
Time Frame: Assessed during surgery and for 30 days after the end of treatment.
Arm/Group | Minimally Invasive Esophagectomy (MIE)
Serious Adverse Events (participants affected / at risk) | 75/105
Other Adverse Events (participants affected / at risk) | 74/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minimally Invasive Esophagectomy (MIE) (N=105)
Anemia (Blood and lymphatic system disorders) | 2
Lymphopenia (Investigations) | 1
Atrial fibrillation (Cardiac disorders) | 3
Cardiac-ischemia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Insomnia (Psychiatric disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
Constitutional, other (General disorders) | 1
PTT (Investigations) | 1
Wound - non-infectious (Injury, poisoning and procedural complications) | 1
Death NOS (General disorders) | 1
Death - multiorgan failure (General disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Dysphagia (Gastrointestinal disorders) | 19
Fistula, Colon/cecum/appendix (Gastrointestinal disorders) | 1
Fistula, Esophageal (Gastrointestinal disorders) | 4
Ileus (Gastrointestinal disorders) | 1
Leak (including anastomotic, esophagitis) (Injury, poisoning and procedural complications) | 10
Nausea (Gastrointestinal disorders) | 3
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1
Obstruction, stomach (Gastrointestinal disorders) | 1
Stenosis (including anastomotic) esophagus (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 2
GI-other (Gastrointestinal disorders) | 6
Hematoma (Vascular disorders) | 2
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 1
Surgical hemorrhage (Injury, poisoning and procedural complications) | 3
Colitis, infectious (e.g. C.diff) (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, jejunum (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, lung (Infections and infestations) | 8
Infection w/ Gr0-2 neutropenia, mediastinm (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, neck NOS (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, pleura (Infections and infestations) | 2
Infection w/ Gr0-2 neutropenia, upper airway (Infections and infestations) | 1
Infectionw/ Gr0-2 neutropenia, wound (Infections and infestations) | 2
Infection w/ unknown ANC foreign body (Infections and infestations) | 1
Infection w/ unknown ANC lung (Infections and infestations) | 4
Infection w/ unknown ANC peritoneal cavity (Infections and infestations) | 1
Infection w/ unknown ANC pleura (empyema) (Infections and infestations) | 1
Infection w/ unknown ANC upper aerodigest (Infections and infestations) | 1
Opportunistic infection lymphopenia>=grade 1 (Infections and infestations) | 1
Infection w/ Gr0-2 neutropenia, blood (Infections and infestations) | 1
Chyle or lymph leakage (Vascular disorders) | 1
Edema limb (General disorders) | 1
Edema trunk/genital (General disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
ALT increased (Investigations) | 1
AST increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Laryngeal nerve dysfunction (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 3
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 2
Esophagus, pain (Gastrointestinal disorders) | 1
Pain NOS (General disorders) | 1
Pleura, pain (General disorders) | 2
Pain-other (General disorders) | 2
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Fistula trachea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Obstruction, airway-larynx (Injury, poisoning and procedural complications) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 14
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Prolong intubation post pulm resection (Injury, poisoning and procedural complications) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2
Intra-op injury Spleen (Injury, poisoning and procedural complications) | 1
Intra-op injury Vein inferior vena cava (Injury, poisoning and procedural complications) | 1
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Minimally Invasive Esophagectomy (MIE) (N=105)
Anemia (Blood and lymphatic system disorders) | 11
Atrial fibrillation (Cardiac disorders) | 14
Dysphagia (Gastrointestinal disorders) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 28
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No